CLINICAL TRIAL: NCT03504527
Title: Effeciency of Budesonide Combined With Formoterol and Tiotropium in the Treatment of Acute Exacerbation of Asthma-chronic Obstructive Pulmonary Overlap: A Randomized Controlled Clinical Study
Brief Title: Efficiency of Budesonide Combined With Formoterol and Tiotropium in the Treatment of Acute Exacerbation of ACO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Shengqing Li, Chief physician, professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2017-008
Record Dates: First submitted 2017-09-28; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Asthma-COPD Overlap
Keywords: ICS; LABA; LAMA; therapy; asthma; COPD; ACO
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- triple combinations (Experimental): Budesonide/Fermotil inhalant 160ug/4.5ug bid; Tiotropium bromide inhalants 18ug qd
  Interventions: Drug: triple combinations
- double combinations (Active Comparator): Fermotil inhalants 4.5ug bid; Tiotropium bromide inhalants 18ug qd
  Interventions: Drug: double combinations

INTERVENTIONS:
Drug: triple combinations — inhaled budesonide(160ug,bid),formotero(4.5ug,bid) and tiotropium bromide(18μg,qd)
  Other Names: budesonide/formotero/tiotropium bromide triple combinations
  Arms: triple combinations
Drug: double combinations — inhaled formotero(4.5ug,bid) and tiotropium bromide(18μg,qd)
  Other Names: formotero/tiotropium bromide double combinations
  Arms: double combinations

SUMMARY:
This study evaluates the efficiency of ICS(budesonide) combined with LABA (formoterol) and LAMA(tiotropium) in the treatment of acute exacerbation of asthma-chronic obstructive pulmonary overlap. Half of participants will receive budesonide,formoterol and tiotropium in combination, while the other half will receive budesonide and formoterol only.

DETAILED DESCRIPTION:
ACO(asthma-chronic obstructive pulmonary overlap) is a relatively new proposed clinical form of chronic airway disease. Guideline or preferring therapy for ACO is still evolving. Current clinical solution is when ACO presents like asthma, initial treatment will accord to the guideline for asthma , while it presents like COPD, COPD recommendation treatment (not alone ICS,but ICS in addition of LABA with or without LAMA) will be chosen, which are subjective. Although present guidelines has recommended that ACO should be treated with at last two inhalant, but limited date have proven it.

A random controlled trial will be conducted to evaluate the efficiency of ICS(budesonide) combined with LABA (formoterol) and LAMA(tiotropium bromide) in the treatment of acute exacerbation of ACO,compared with the control group receiving tiotropium bromide with formoterol only.

ELIGIBILITY:
Inclusion Criteria:

* subject has ACO

Exclusion Criteria:

* acute exacerbation of ACO;
* acute infection;
* postbrochodilator FEV1/FVC> 0.7;
* pulmonary complications: bronchiectasis, active tuberculosis, pulmonary fungal disease or lung cancer
* history of other malignant tumor
* with rheumatic diseases;
* with some serious heart, cerebrovascular, liver, kidney or hematopoietic system diseases
* with tachyarrhythmias；
* mental patients;
* with moderate to severe renal insufficiency (creatinine clearance ≤ 50ml / h)
* allergic to the budesonide, formoterol or tiotropium bromide;
* history of acute gastrointestinal bleeding within 3 months;
* with severe angle closure glaucoma patients;
* pregnancy,lactation;
* have participated in other clinical trials in 3 months；
* hospital staff and their relatives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
the frequency of ACO exacerbation | 12 months
  the frequency of ACO exacerbation

SECONDARY OUTCOMES:
postbronchodilator FEV1 | 12 months
  a post-bronchodilator forced expiratory volume in one second
times of hospital readmission caused by exacerbation | 12 months
  times of hospital readmission caused by exacerbation
other lung function parameters | 12 months
  other lung function parameters(%FEV1, FEV1/FVC)
CCQ score | 12 months
  Clinical COPD Questionnaire score
mMRC score | 12 months
  modified Medical Research Council score
CAT score | 12 months
  COPD Assessment Test score
ACT score | 12 months
  Asthma Control Test score

CONTACTS AND LOCATIONS:
Overall Officials: Li Shengqing, PhD, Principal Investigator — Huashan Hospital

IPD SHARING:
Plan to Share IPD: No